CLINICAL TRIAL: NCT02766764
Title: Evaluation of the Role of Combined Dehydropeiandrosterone and Growth Hormone in Women With Expected Poor Ovarian Response Undergoing ICSI: A Double Blind Placebo Controlled Study.
Brief Title: Combined Dehydropeiandrosterone and Growth Hormone in Women With Expected Poor Ovarian Response Undergoing ICSI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DHEA 4
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Subfertility
MeSH Terms: conditions — Infertility | interventions — Dehydroepiandrosterone; Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (Active Comparator): Women will receive oral DHEA 25 mg t.d.s daily for 12 weeks before ICSI in addition to daily GH injections from day 6 of hMG administration until the day of hCG administration.
  Interventions: Drug: DHEA; Drug: Growth hormone
- Placebo group (Placebo Comparator): Women will receive an oral placebo similar to DHEA t.d.s daily for 12 weeks before ICSI in addition to daily placebo injections similar to GH from day 6 of hMG administration until the day of hCG administration.
  Interventions: Drug: Placebo 1; Drug: Placebo 2

INTERVENTIONS:
Drug: DHEA — Women will receive oral DHEA 25 mg t.d.s. for 12 weeks before ICSI.
  Arms: Study group
Drug: Growth hormone — Women will receive GH subcutaneous injections daily from day 6 of hMG administration until the day of hCG administration.
  Arms: Study group
Drug: Placebo 1 — Women will receive an oral placebo similar to DHEA t.d.s for 12 weeks before ICSI
  Arms: Placebo group
Drug: Placebo 2 — Women will receive subcutaneous placebo injections similar to GH daily starting from day 6 of hMG injections until the day of hCG injection
  Arms: Placebo group

SUMMARY:
Two hundred and thirty women with expected poor ovarian response undergoing IVF/ICSI will be randomly divided into 2 equal groups using computer generated random numbers. Group 1 will receive DHEA 25 mg (DHEA 25mg, Natrol , USA) t.d.s for 12 weeks before starting IVF/ICSI cycle in addition to Growth hormone (GH; Somatotropin, Sedico, Egypt) 4 IU on day 6 of human menopausal gonadotropin (hMG) stimulation in a daily dose of 2.5 mg subcutaneous (sc) until the day of human chorionic gonadotropin (hCG) triggering Group 2 will receive an oral placebo t.d.s. daily for 12 weeks before ICSI in addition to a sc placebo similar to GH daily from day 6 of stimulation until the day of hCG trigger.

DETAILED DESCRIPTION:
The study will be conducted in Cairo university hospitals and Dar Al-Teb Infertility and Assisted conception center, Giza Egypt. All patients will be evaluated for their expected ovarian response. Patients fulfilling the Bologna criteria definition of poor ovarian response will be invited to participate in the study and to sign informed consent forms.

Two hundred and thirty women with expected poor ovarian response (POR) undergoing IVF/ICSI will be randomly divided into 2 equal groups using computer generated random numbers. Group 1 will receive DHEA 25 mg (DHEA 25mg, Natrol , USA) t.d.s daily for 12 weeks before starting IVF/ICSI cycle in addition to GH Growth hormone (Somatotropin, Sedico, Egypt) 4 IU on day 6 of hMG stimulation in a daily dose of 2.5 mg SC until the day of hCG triggering Group 2 will receive an oral placebo t.d.s. daily for 12 weeks before ICSI in addition to a placebo similar to GH daily from day 6 of stimulation until the day of hCG trigger.

Patients included in the study will be subjected to full history taking and clinical examination. On the second day of menstruation serum FSH, LH, Prolactin and Oestradiol will be assessed and the antral follicular count (AFC) will be assessed using a vaginal ultrasound scan. AFC will be defined as the number of follicles measuring 3-10mm.

All patients will have gonadotropin antagonist protocol with Human menopausal gonadotrophin (HMG) stimulation until the day of (Human chorionic gonadotrophin (HCG) administration. On the second day of menstruation serum FSH, LH, Prolactin and Oestradiol will be assessed and the antral follicular count (AFC) will be assessed using a vaginal ultrasound scan. AFC will be defined as the number of follicles measuring 3-10mm.

The stimulation protocol will start on day 2 using 450-300 IU HMG ( Merional® IBSA, Lugano, Switzerland) and GnRH antagonist, cetrorelix (Cetrotide® Merck Serono, Darmstadt, Germany) 0.025 mg daily. Gonadotropins will be administered for 4 to 5 days, after which the dose will be adjusted according to the ovarian response. The ovarian response will be monitored by transvaginal ultrasound and serum E2 levels. When three or more follicles reached a maximum diameter of 16 mm, highly purified HCG 5000 or 10,000 IU (Choriomon ®IBSA) will be administered. The procedure will be cancelled if less than 3 follicles 16 mm in size are present 12 days after starting gonadotropins despite doses reaching 450 IU. The cycle will be also cancelled if there is risk of ovarian hyperstimulation like massive ovarian enlargement or serum estradiol exceeds 3000pg/L Transvaginal oocyte retrieval will be performed 34-36 h after the administration of HCG. Oocytes will be fertilized either via IVF or ICSI based on the couple's history. Fertilization will be assessed 16-18 h after IVF or ICSI. Embryos will be transferred on Day 3 or 5. Vaginal tablets containing progesterone (Prontogest® IBSA) 400 mg/day will be given when fertilization is confirmed. A pregnancy test will be done 2 weeks after embryo transfer. For patients with a positive pregnancy test, progesterone is to be continued for an additional 4 weeks. Clinical pregnancy will be defined as Visualization of an intrauterine gestational sac 5 weeks after embryo transfer. And ongoing pregnancy will be defined as the sonographic confirmation of fetal heart pulsations at 12 weeks.

Sample size calculation:

The researchers are planning a study of independent cases and controls with 1 control(s) per case. Kotb et al found that the ongoing pregnancy rate in women undergoing IVF/ICSI who received DHEA with expected POR according to the Bologna criteria is 0.285 versus 0.128 in the control group. Assuming that adding GH to DHEA will not increase the ongoing pregnancy rate, the researchers will need to study 103 case patients and 103 control patients to be able to reject the null hypothesis that the exposure rates for case and controls are equal with probability (power) 0.8. The researchers added 12 patients to each arm accounting for any missing data or losses to follow up. The Type I error probability associated with this test of this null hypothesis is 0.05. The researchers used an uncorrected chi-squared statistic to evaluate this null hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing ICSI with expected poor ovarian response according to the Bologna criteria

Exclusion Criteria:

* Body mass index >35 Kg/m2.
* Women with a single ovary.
* Allergy to DHEA or GH.
* Diabetic women on insulin as insulin lowers DHEA levels and might reduce its effectiveness

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 230 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy | 12 weeks after embryo transfer
  Ongoing pregnancy will be defined as the confirmation of fetal heart pulsations using trans-vaginal ultrasound 12 weeks after embryo transfer.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Cairo university hospitals, Cairo
  - Dar AlTeb subfertility centre, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kotb MM, Hassan AM, AwadAllah AM. Does dehydroepiandrosterone improve pregnancy rate in women undergoing IVF/ICSI with expected poor ovarian response according to the Bologna criteria? A randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2016 May;200:11-5. doi: 10.1016/j.ejogrb.2016.02.009. Epub 2016 Feb 21. PMID 26963897
- [Background] Bassiouny YA, Dakhly DMR, Bayoumi YA, Hashish NM. Does the addition of growth hormone to the in vitro fertilization/intracytoplasmic sperm injection antagonist protocol improve outcomes in poor responders? A randomized, controlled trial. Fertil Steril. 2016 Mar;105(3):697-702. doi: 10.1016/j.fertnstert.2015.11.026. Epub 2015 Dec 13. PMID 26690008
- [Background] Dakhly DM, Bayoumi YA, Gad Allah SH. Which is the best IVF/ICSI protocol to be used in poor responders receiving growth hormone as an adjuvant treatment? A prospective randomized trial. Gynecol Endocrinol. 2016;32(2):116-9. doi: 10.3109/09513590.2015.1092136. Epub 2015 Sep 29. PMID 26416521
- [Background] Bayoumi YA, Dakhly DM, Bassiouny YA, Hashish NM. Addition of growth hormone to the microflare stimulation protocol among women with poor ovarian response. Int J Gynaecol Obstet. 2015 Dec;131(3):305-8. doi: 10.1016/j.ijgo.2015.05.034. Epub 2015 Aug 23. PMID 26381201